CLINICAL TRIAL: NCT02828787
Title: Central Mechanisms of Chronic Pruritus: Functional and Structural Brain Imaging.
Acronym: PRURIM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of the inclusion period. A late start of inclusions and reduced scanner availability meant that the number of 45 participants could not be reached.
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RB 15.212 PRURIM
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Urticaria (Experimental): 15 patients with urticaria
  Interventions: Other: MRI
- Psoriasis (Experimental): 15 patients with psoriasis
  Interventions: Other: MRI
- healthy (Other): 15 healthy control subjects
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — The study will take place in two phases. The first phase consists of a meeting of inclusion. During this phase, the principal investigator of the study will verify the inclusion criteria for patients using a questionnaire and an interview. Then, the effects of video on each person will be tested to verify that they well induce itch and measure it using visual analogue scales. This phase will also test the benefit of the relief by scraping and cold.
  The second phase will be carried out only if the mental induction of pruritus has been possible in the first session. It involves acquiring the corresponding physiological signals fMRI. It will also be achieved during this phase an anatomical image of the brain of each participant and an image in DTI.
  The phases will be carried out in this order in each participant. They will be separated at least one night.

SUMMARY:
The main objective of this study is to identify by functional and structural MRI which are the brain areas activated in various pruritic situations to deduct a model describing the different causes of pruritus.

The investigators are going to compare two chronic pruritus conditions (histaminergic urticaria and non histaminergic: psoriasis) to a healthy control group.

The secondary objective of this study is to specify a classification index from the physiological results obtained by brain imaging to differentiate multiple types of pruritus.

DETAILED DESCRIPTION:
Particularly invalidating in some cases, pruritus is defined as an unpleasant sensation that causes the need to scratch.

Epidemiologically, it is a common disorder as a third of the population feels in a given week. Treatment is difficult, especially as the pathophysiological mechanisms remain poorly understood, particularly in the central nervous system.

Specific pathways, or at least selective of the pruritus of transmission have been identified. From the skin to the brain, two ways exist: a histaminergic pathway (classical), and a non-histaminergic pathway (related to the activation of PAR-2 receptors by serine proteases). If urticaria belongs to the first track, the respective share of each channel is unknown to other causes of pruritus. The pruriceptors, located in the skin, transmit information by specific fibers at the spinal cord, which then project through the lateral spinothalamic tract to the thalamus. Then at midbrain and cortex, a vast network involving sensorial areas, motor and emotional areas was identified by functional neuroimaging, with activation zones which may be different depending on two channels (with overlapping zones ). The contribution to the perception of pruritus of these brain regions is the focus of current research.

A promising non-invasive method to study the pruritus channels with neuroimaging is to use the phenomenon of "contagious pruritus': seeing other people scratching, itching and sometimes scratching is induced in the observer, and the activated brain network is similar to that which is activated by pruritus usually. This phenomenon is even more important in subjects with atopic dermatitis than in healthy subjects.

In this project, the investigators plan to characterize pruritus central pathways in patients with different types of chronic pruritus compared to healthy subjects, particularly regarding the respective contributions of histaminergic pathways (pathway involved in pruritus of hives) and "PAR-2-ergic" (pathway involved in the itch of psoriasis).

ELIGIBILITY:
Inclusion Criteria:

* Or patient affected by psoriasis presenting a pruritus of more than 6 weeks
* Or patient affected by urticaria presenting a pruritus of more than 6 weeks
* Or subject without dermatosis and not presenting chronic pruritus.
* Major
* Able to provide written informed consent
* Affiliated to the Social Security

Exclusion Criteria:

1. In connection with the award of an MRI namely:

   * The presence of implanted medical equipment susceptible to the magnetic field of MRI,
   * Claustrophobia
   * Medication, treatment and / or substances that could alter or modify brain function
   * Pregnancy
2. In connection with the mode of presentation of stimuli (video):

   - An uncorrected visual disorder not allowing to view videos
3. In connection with the administrative regulations:

   * Persons under 18
   * Major Persons subject to legal protection (backup justice, trusteeship, guardianship), persons deprived of liberty.

If no pruritus is induced during the first session, it will be a criterion for non inclusion for the second session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
brain areas activated during a mentally induced pruritus in 3 different populations | 1 year
  The primary endpoint is to highlight fMRI brain areas activated during a mentally induced pruritus in 3 different populations: healthy subjects (no pre-existing pruritus), patients with chronic urticaria (pruritus related to histaminergic pathway), and psoriasis patients (activation pathway pruritus probably PAR2-ergic but to be confirmed by the study).

SECONDARY OUTCOMES:
index, form the combination the better able to explain the membership of an individual (individual analysis) to a pathological community or not. | 1 year
  The secondary outcome is to verify that data collected, once grouped and established in index, form the combination the better able to explain the membership of an individual (individual analysis) to a pathological community or not.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Laurent MISERY, Brest
  - CHRU de Brest, Brest

IPD SHARING:
Plan to Share IPD: No